CLINICAL TRIAL: NCT04786821
Title: Feasibility Study for a Randomised Control Trial for the Acceptability of Exoskeleton Assisted Walking Compared to Standard Exercise Training for Persons With Mobility Issues Due to Multiple Sclerosis
Brief Title: Acceptability of Exoskeleton Assisted Walking for Persons With Mobility Issues Due to Multiple Sclerosis
Acronym: ExoMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STH20833
Record Dates: First submitted 2021-01-18; First posted 2021-03-08 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; Pathologic Processes; Sclerosis; Autoimmune Diseases of the Nervous System; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases
Keywords: Exoskeleton Device; Exercise Programme
MeSH Terms: conditions — Multiple Sclerosis; Pathologic Processes; Sclerosis; Autoimmune Diseases of the Nervous System; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: The eligible participants will be allocated to either arm using an online randomisation site in 1:1 randomisation ratio. All participants will have equal chance of getting allocated to either arm.
Who Masked: Outcomes Assessor
Masking Description: It is not practical to blind the participants to the intervention as the study team are studying two different types of physical activities. The study team will explore whether it is feasible for the outcome assessor to be blind to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Exercise Training Programme (Placebo Comparator): Participants will receive interventions by an exercise specialist based on the participant's tolerance. These sessions will be delivered by a exercise specialist.
  Interventions: Behavioral: Standard Exercise Training
- Exoskeleton Exercise Programme (Active Comparator): The Phoenix Exoskeleton suit will be used in this study. It is a powered Exoskeleton, with a modular design. Participants will receive interventions by an research physiotherapist based on the participant's tolerance.
  Interventions: Device: Phoenix Exoskeleton suit

INTERVENTIONS:
Behavioral: Standard Exercise Training — Participants will receive interventions by an exercise specialist for up to 30 minutes based on the participant's tolerance. The exercises used in control group will depend on the individual and their abilities as evaluated in the baseline assessment session. Possible exercises include arm crank, recumbent cycle, and chair exercises. These sessions will be delivered by a member of the research team.
  Arms: Standard Exercise Training Programme
Device: Phoenix Exoskeleton suit — Participants will aim to walk wearing the Exoskeleton for up to 30 minutes. Based on the participant's tolerance, the duration of walking can be shorter and can be split into shorter intervals to achieve more activity. Over the sessions, based on the participants' tolerance, gradually the duration of walking can be increased with shorter breaks. This will be delivered by a research physiotherapist.
  Arms: Exoskeleton Exercise Programme

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory disease of the central nervous system. Lack of physical activity is common in people with MS (pwMS). This can lead to several comorbid conditions such as obesity, metabolic syndrome, osteoporosis, hypertension, diabetes and worse prognosis. An increasing number of studies suggest that physical exercise can play an important role in managing symptoms, preventing complications and comorbidities in pwMS, and may possibly be neuroprotective. However, doing exercise can be very challenging for pwMS who have moderate/severe mobility disability and who have problems with walking.

In this project, the investigators will explore the use of a powered Exoskeleton as an exercise tool for people with moderate to severe difficulty walking due to MS. Powered Exoskeletons are wearable robots that offer opportunity to persons with lower limb weakness to stand and walk. The Exoskeleton-assisted training provides active training with potentially much less intervention needed from therapists. However, it is not clear whether pwMS can walk with a powered Exoskeleton at speeds and intensities sufficient to positively affect health and fitness outcomes. Thus, in this study, the investigators aim to explore whether using an Exoskeleton will enable people with MS to exercise at a moderate intensity and whether people with MS find this acceptable and safe to do on a regular basis. The investigators will also explore whether training with an Exoskeleton can improve walking. The investigators will train 12 patients with MS to walk with an Exoskeleton twice a week for 8 weeks. The investigators will compare the effects with another group of 12 patients who will do exercises with a fitness instructor twice a week for 8 weeks. The investigators will study whether walking with Exoskeleton is better than fitness training in terms of fitness outcomes, walking and cognitive, psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS as per the McDonald criteria (Polman et al., 2011).
* Age 18 years or older.
* Cognitive ability to give consent and participate in the protocol.
* Walking limitations with Expanded Disability Status Scale (EDSS) scores ranging from 5.0 to 7.5.
* Enough strength in hands and shoulders to support themselves standing and walking using crutches or a walker.
* Meet the general requirements to fit with the Phoenix Exoskeleton (160-190.5 cm in height, weight below 80 Kg, hip width no greater than 42.7 cm measured when sitting, healthy skin where it touches Phoenix Exoskeleton).
* Able to tolerate exercise twice per week as judged by the PI during screening.

Exclusion Criteria:

* Any illness, other than MS, affecting walking and exercise performance.
* Severe cognitive or behavioral impairment.
* Relapses 3 months prior to enrolment.
* Change in disease modifying drugs for MS 6 months before enrolment.
* Botulin toxin injections for the lower limbs the previous 3 months.
* Any medical contraindications to assisted walking (e.g., cardiovascular condition, weight-bearing restrictions, osteoporosis or other fracture risk, pregnancy, uncontrolled seizure).
* Significant flexion contractures limited to 35 degrees at the hip and 20 degrees at the knee that precluded Phoenix Exoskeleton fit.
* Psychopathology or other health conditions that the physiotherapist, in his or her clinical judgement, considers to be exclusionary to safely use an Exoskeleton.
* Living more than 20 miles away from the experiment location to reduce burden on patients due to the number of planned study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate estimation | One day
  The research team will identify the number of potential participants who responded to our initial recruitment strategies and the proportion who remain interested after being informed of the requirements of the study. Feasibility will be classed as 60% or more of eligible participants consenting to the trial.
Retention rate estimation | 8 weeks
  Adherence will be measured through attendance at the Exoskeleton and exercise sessions and compliance to the protocol. Feasibility will be classed as 75% of the recruited participants completing 12 or more of the 16 intervention sessions (not including the familiarisation sessions). Patient Participation will be assessed by the research physiotherapist and exercise therapist using the Pittsburg Participation Questionnaire.
Acceptability of the intervention - VAS | 8 weeks
  Data from participant's visual analogue scale of patient discomfort will be used to determine acceptability. Feasibility will be defined as less than 1/3 of participants reporting moderate or greater discomfort on the visual analogue scale. Throughout the study, participants asked to score discomfort experienced on VAS scale 0-10 where 0=no discomfort and 10=intolerable.
Acceptability of the intervention - Patient perception questionnaire | 8 weeks
  A patient perception questionnaire will be used to gather more in-depth qualitative data about acceptability. This will give us insight into the acceptability of the type of exercise and any benefits that have been derived, helping us to take the project forward in the future and design an intervention that fits with the requirements of this population group.

SECONDARY OUTCOMES:
Number of participants achieving target heart rate | 8 weeks
  Heart rate will be monitored throughout the intervention sessions. This will be used to explore the level of exercise stimulation achieved through powered exoskeleton walking compared to exercise training.
Aerobic Fitness (arm cranking) | 8 weeks
  To be completed at baseline and follow up. This will be used to explore the level of exercise stimulation achieved through powered exoskeleton walking compared to exercise training.
Waist to hip ratio | 8 weeks
  Waist to hip ratio measurement is calculated by dividing the measurement of the waist by the hip measurement. To be completed at baseline and follow up.
Body fat percentages | 8 weeks
  Body fat percentage, measures a person's relative body composition without regard to height or weight. To be completed at baseline and follow up.
10 metre walking gait test wearing inertial sensors | 8 weeks
  This will only be completed in participants that are able to walk minimum of 2 metres with or without assistance. To be completed at baseline and follow up. To assess the effect of Exoskeleton and exercise training on gait.
Multiple Sclerosis Impact Scale (MSIS-29) | 8 weeks
  Multiple Sclerosis Impact Scale (MSIS-29) used to capture views about the impact of MS on participants day-to-day life during the past two weeks. To be completed at baseline and follow up to assess the impact of Exoskeleton and exercise training on MS related symptoms and quality of life. MSIS-29 provides a score between 29-145 where larger scores indicate that MS has a greater impact on day-to-day life for the participant.
Modified Fatigue Impact Scale (MFIS) | 8 weeks
  Modified Fatigue Impact Scale (MFIS) will be used to assess how fatigue impacts individuals lives in the past 4 weeks. To be completed at baseline and follow up to assess the impact of Exoskeleton and exercise training on MS related symptoms and quality of life.. Scores range between 0-84 where larger scores indicate greater impact of fatigue on daily life.
Multiple Sclerosis walking scale (MSWS-12) | 8 weeks
  Multiple Sclerosis walking scale (MSWS-12) used to capture a self-reported measure of the impact of MS on the individual's walking ability in the past 2 weeks. To be completed at baseline and follow up to assess the impact of Exoskeleton and exercise training on MS related symptoms and quality of life. Scores range between 12-60 where larger scores indicate greater impact of MS on walking activities.
The Borg rating of perceived exertion scale | 8 weeks
  Participant's will be asked to rate physical activity intensity level throughout the study. Borg RPE scale will be used, 6-20 where 6 = no effort at all and 20= absolute maximal effort. This will be used to explore the level of exercise stimulation achieved through powered Exoskeleton walking compared to exercise training.
Quality of life questionnaire (EQ-5D-5L & VAS) | 8 weeks
  EuroQol quality of life questionnaire (EQ-5D-5L) will be used to capture views about the participants quality of life within 24hours in 5 themes. Using the VAS scores, participants will rate their quality of life between 100 = the best health you can imagine and 0 = the worst health you can imagine. To be completed at baseline and follow up. This will be used to assess the impact of Exoskeleton and exercise training on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Krishnan Padmakumari Sivaraman Nair, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust; Anouska Carter, Study Chair — Sheffield Hallam University; Christine Smith, Study Director — Sheffield Hallam University
Locations (1):
- sheffield teching hospital NHS foundation trust, Sheffield, South Yorkshire, United Kingdom